CLINICAL TRIAL: NCT05590494
Title: Ultrasonic Tenotomy as a Treatment of Partial Rotator Cuff Tear of the Supraspinatus Tendon: A Pilot Feasibility Study
Brief Title: Novel Treatment for Rotator Cuff Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jacob L. Erickson, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-011522
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Supraspinatus Tear
Keywords: Ultrasonic tenotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Repair a partially torn rotator cuff (Other): Subjects will undergo an ultrasonic tenotomy to repair a partially torn rotator cuff per standard of care as clinically indicated
  Interventions: Procedure: Ultrasonic tenotomy

INTERVENTIONS:
Procedure: Ultrasonic tenotomy — Ultrasonic procedure as part of standard of care, as clinically indicated, to stimulate healing of the partial tear. The procedure uses ultrasound guidance that allows a needlelike device to gradually break up and remove tendinopathic tendon tissue.

SUMMARY:
The focus of this study is to examine changes in pain scores, strength, and range of motion over time following an ultrasonic tenotomy on a partial tear (<50%) of the supraspinatus tendon of the rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

- Evidence of partial tear (< 50%) of the supraspinatus tendon on MRI.

Exclusion Criteria:

* A tear of the supraspinatus tendon greater > 50% and any areas of full thickness tearing, concomitant tears > 25% of other rotator cuff tendons (infraspinatus, teres minor or subscapularis), or acute tear of the glenoid labrum.
* Evidence of systemic illness/infection requiring oral or IV antibiotics during the recruitment period.
* Evidence of overlying skin infection or lesion at the proposed device insertion point on the shoulder.
* Previous corticosteroid injection within three months.
* Those individuals less than 25 and greater than 75 years of age will be excluded.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain | Baseline, 2, 6, 12 and 24-weeks post-procedure
  Measured using a visual analog scale (VAS), used to measure subjective pain, rated from 0 (no pain) to 100 (most severe pain) at rest and during activity (previously painful activities)
Change in shoulder active range of motion | Baseline, 2, 6, 12 and 24-weeks post-procedure
  Measured using a goniometer reported in degrees
Change in shoulder strength | Baseline, 2, 6, 12 and 24-weeks post-procedure
  Assessed using a hand-held dynamometer (HHD) placed distally on the forearm, just proximal to the wrist joint along the distal radius and ulna with instruction to push into the HHD with maximum force production for approximately 5 seconds.

SECONDARY OUTCOMES:
Change in quality of life | Baseline, 2, 6, 12 and 24-weeks post-procedure
  Measured using the SF-36 Quality of Life questionnaire which is a 36-item self-reported health survey that measures health and disability. Possible scores range from 0 to 100, with 0 indicating maximum disability, and 100 indicating no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Erickson, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System - Onalaska, Onalaska, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials